CLINICAL TRIAL: NCT05710692
Title: A Multicenter Open-Label Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of Pegunigalsidase Alfa (PRX-102) in Japanese Patients With Fabry Disease (RISE)
Brief Title: Study to Evaluate the Safety, PK, PD, and Efficacy of PRX-102 in Japanese Patients With Fabry Disease
Acronym: RISE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-06657AA2-01
Record Dates: First submitted 2022-12-13; First posted 2023-02-02 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRX-102 1 mg/kg every 2 weeks or PRX-102 2 mg/kg every 4 weeks (Experimental): PRX-102 1 mg/kg every 2 weeks or PRX-102 2 mg/kg every 4 weeks (available only in the optional extension part)
  Interventions: Drug: PRX-102 1 mg/kg every 2 weeks; Drug: PRX-102 2 mg/kg every 4 weeks

INTERVENTIONS:
Drug: PRX-102 1 mg/kg every 2 weeks — PRX-102 1 mg/kg every 2 weeks
  Other Names: pegunigalsidase alfa; Recombinant human alpha galactosidase-A
Drug: PRX-102 2 mg/kg every 4 weeks — PRX-102 2 mg/kg every 4 weeks
  Other Names: pegunigalsidase alfa; Recombinant human alpha galactosidase-A

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of pegunigalsidase alfa in Japanese patients (adults and adolescents) affected by Fabry disease. It is planned of a total of approximately 18-20 male and female Fabry disease patients between the ages of 13 and 60 years to be part of the study. The study is conducted in Japan.

DETAILED DESCRIPTION:
Investigators are doing this study to find out if treatment with pegunigalsidase alfa will prevent or reduce the development of health problems caused by Fabry disease and thereby improve patients' health and quality of life.

pegunigalsidase alfa (PRX-102) is a drug made using genetic engineering techniques and manufactured using cultured tobacco cells. It is given by intravenous infusion every 2 weeks, at a dosage of 1 milligram per kilogram (mg/kg) of body weight.

The study consists of a main study that is divided into two stages, each of which will last one year, followed by an optional extension study. In the optional extension stage, the participants may receive PRX-102 intravenous infusion every 2 weeks, at a dosage of 1 milligram per kilogram (mg/kg) of body weight or every 4 weeks at a dosage of 2 milligrams per kilogram (mg/kg) of body weight.

There are three groups (cohorts) in this study, with adults enrolled in either Cohort A or B and adolescents in Cohort C. Whether an adult is assigned to Cohort A or Cohort B depends on their kidney function and treatment history.

This study will start with a screening visit of up to 4 weeks. It will be followed up by infusion visits every 2 weeks or 4 weeks. For subjects not continuing in the extension stage, a follow-up call is to be made 30 days after the last study drug infusion.

ELIGIBILITY:
Inclusion criteria (all subjects)

1. Must have been born in Japan and have their biological parents and all 4 grandparents of Japanese descent
2. A documented diagnosis of Fabry disease, as determined by the following:

   * Males: Plasma and/or leukocyte alpha-galactosidase-A activity (by activity assay) that is ≤ 5% of mean normal laboratory levels or, if the enzymatic activity is above the 5% limit but still under the normal level, a confirmed disease-causing mutation of the GLA gene
   * Females: Historical genetic test results consistent with Fabry mutations or, in the case of novel mutations, a first-degree male relative with Fabry disease
   * All subjects: At least one of the following characteristic features of Fabry disease: neuropathic pain, cornea verticillata, and/or clustered angiokeratoma
3. Estimated glomerular filtration rate (eGFR) at screening ≥40 mL/min/1.73 m2. For adults, this will be calculated using the Japanese Modified Chronic Kidney Disease Epidemiology Collaboration (JPN-CKD-EPI) Creatinine equation (2009); and for adolescents, it will be calculated using the Creatinine Cystatin C-based Chronic Kidney Disease in Children (CKiD) equation.
4. Clinical condition that in the opinion of the Investigator requires treatment with ERT
5. A female subject (including an adolescent in Cohort C, if applicable) must meet one of the following criteria:

   * If of childbearing potential, she must:

     * Have a negative serum pregnancy test result at screening, AND
     * Agree to undergo a urine pregnancy test at baseline and every 12 weeks thereafter up to the final treatment, AND
     * Agree to use one of the following highly reliable methods of contraception from the day of the informed consent signature until 30 days after the last infusion received. The following methods are acceptable:

       * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
       * Combined (both oestrogen and progestogen) hormonal contraception (oral) associated with inhibition of ovulation, supplemented with a barrier method (preferably male condom)
       * Bilateral tubal occlusion
       * Sexual abstinence, defined as refraining from heterosexual intercourse during the entire study period
       * Partner vasectomy, provided that the partner is the sole sexual partner and has received medical verification of the surgical success
   * Be of non-childbearing potential, defined as one of the following:

     * Post-menopausal (12 consecutive months of amenorrhea), OR
     * Permanently sterile following hysterectomy, bilateral salpingectomy, or bilateral oophorectomy (supporting evidence required)

Additional inclusion criteria for subjects in Cohort A

For subjects enrolled in Cohort A, these specific inclusion criteria, in addition to those above, apply:

* Aged ≥18 to ≤70 years
* Treatment with agalsidase beta or agalsidase alfa for at least the last 12 months prior to screening, with the dose stable (defined as having received at least 80% of the labelled dose) for at least the last 6 months
* Diagnosis of kidney impairment, defined as a linear slope of eGFR more negative than or equal to -2 mL/min/1.73 m2/year. The historical eGFR slope will be calculated based on at least 3 serum creatinine values obtained over the 9 to 24 months prior to screening, using the JPN-CKD-EPI Creatinine equation (2009). This criterion will be confirmed at screening by calculating the screening eGFR slope using historical and screening serum creatinine values. Both historical and screening eGFR slopes will be used for the diagnosis of kidney impairment.

Additional inclusion criterion for subjects in Cohort B

For subjects enrolled in Cohort B, this specific inclusion criterion, in addition to those above, applies:

- Aged ≥18 to ≤70 years

Additional inclusion criteria for subjects in Cohort C

For subjects enrolled in Cohort C, these specific inclusion criteria, in addition to those above, apply:

* Aged ≥13 to <18 years
* Subjects who have previously received or are currently receiving ERT treatment, must be negative for ADAs to PRX-102

Exclusion Criteria:

1. Administration of ERT for Fabry disease within 14 days before baseline, substrate reduction therapy for Fabry disease within 3 days before baseline, or chaperone therapy for Fabry disease within 3 days before baseline
2. History of type I hypersensitivity reactions (anaphylactic or anaphylactoid life-threatening reaction) to other ERT treatment for Fabry disease or to any component of the study drug
3. Cohort A only: eGFR value of >90 to ≤120 mL/min/1.73 m2 at screening and a historical eGFR value >120 mL/min/1.73 m2 in the 9 to 24 months before screening, indicating absence of renal impairment. eGFR to be calculated using the JPN-CKD-EPI creatinine equation (2009).
4. Urine protein to creatinine ratio (UPCR) >0.5 g/g (0.5 mg/mg or 500 mg/g) if not treated with an ACE inhibitor or ARB
5. Initiation of treatment, or a change in dose to ongoing treatment, with an angiotensin-converting-enzyme inhibitor (ACEI) or angiotensin II receptor blocker (ARB) in the 4 weeks prior to screening.
6. Currently taking another investigational drug for any condition
7. Carry only known non-pathogenic Fabry mutations
8. History of renal dialysis or kidney transplantation
9. History of acute kidney injury in the 12 months prior to screening, including specific kidney diseases (e.g., acute interstitial nephritis, acute glomerular and renal vasculitis); non-specific conditions (e.g., ischemia, toxic injury); or extrarenal pathology (e.g., prerenal azotaemia, and acute postrenal obstructive nephropathy
10. History of (or current) malignancy requiring treatment; the one exception is a prior history of resected basal cell carcinoma
11. Severe cardiomyopathy or significant unstable cardiac disease within 6 months prior to screening
12. A positive test for Severe Acute Respiratory Syndrome-Coronavirus 2 (SARS-CoV-2) within 3 months prior to screening, using a validated molecular assay or validated antigen assay
13. Females: Pregnant or lactating, or of childbearing potential with a fertile male partner and unwilling to use a highly reliable method of contraception from the informed consent signature until 30 days after the last infusion received
14. Presence of any medical, emotional, behaevioral, or psychological condition that in the judgment of the Investigator could interfere with the subject's compliance with the requirements of the study
15. Previous treatment with cellular therapy or gene therapy for any condition

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Incidence of Infusion Related Reactions (IRRs) | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Incidence of Injection site reactions (ISRs) | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change of laboratory tests' results | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change in in body weight in kilograms | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change in height in centimeters | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change in Tanner stage | 12 Months, 24 Months and through study completion (an average of 4.5 years)
  Tanner Staging of Sexual Development will be used to assess sexual development (i.e. breast development (B1 to B5) and pubic hair development (Ph-1 to Ph-5) in females and pubic hair and genetical development (G1-G5) in males.
Change from baseline of 12-lead ECG quantitative parameters: Mean Heart Rate, PR Interval, QRS Duration, QT Interval, QTc Interval, and ST Segment | 12 Months, 24 Months and through study completion (an average of 4.5 years)
  Quantitative ECG parameters will be summarized by cohort and overall
Incidence of treatment-emergent Anti-Drug Antibodies (ADAs) | 12 Months, 24 Months and through study completion (an average of 4.5 years)
ADA status change from baseline | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Incidence of premedication use at each visit and change of infusion premedications from baseline | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change from baseline of Maximum plasma concentration (Cmax), pharmacokinetic parameter | Assessments will be done over three two-week periods, starting at Baseline (Week 0), V7 (Week 12), and V27 (Week 52)
Change from baseline of Time to maximum plasma concentration (tmax), pharmacokinetic parameter | Assessments will be done over three two-week periods, starting at Baseline (Week 0), V7 (Week 12), and V27 (Week 52)
Change from baseline of Area under the plasma concentration-time curve from time 0 to time t (AUC0 t), pharmacokinetic parameter | Assessments will be done over three two-week periods, starting at Baseline (Week 0), V7 (Week 12), and V27 (Week 52)
Change from baseline of Area under the curve from time 0 to 2 weeks (AUC0-2wk), pharmacokinetic parameter | Assessments will be done over three two-week periods, starting at Baseline (Week 0), V7 (Week 12), and V27 (Week 52)
Change from baseline of Area under the curve from time 0 to infinity (AUC0-∞), pharmacokinetic parameter | Assessments will be done over three two-week periods, starting at Baseline (Week 0), V7 (Week 12), and V27 (Week 52)
Change from baseline of Terminal half-life (t1/2), pharmacokinetic parameter | Assessments will be done over three two-week periods, starting at Baseline (Week 0), V7 (Week 12), and V27 (Week 52)
Change from baseline of Area under the curve over a dosing interval (AUCτ), pharmacokinetic parameter | Assessments will be done over three two-week periods, starting at Baseline (Week 0), V7 (Week 12), and V27 (Week 52)
Change from baseline of Observed drug concentration at the end of the dosing interval (Cτ), pharmacokinetic parameter | Assessments will be done over three two-week periods, starting at Baseline (Week 0), V7 (Week 12), and V27 (Week 52)
Change from baseline of Clearance (Cl), pharmacokinetic parameter | Assessments will be done over three two-week periods, starting at Baseline (Week 0), V7 (Week 12), and V27 (Week 52)
Change from baseline of Volume of distribution (Vz), pharmacokinetic parameters | Assessments will be done over three two-week periods, starting at Baseline (Week 0), V7 (Week 12), and V27 (Week 52)

OTHER OUTCOMES:
Change in eGFR | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change in annualized eGFR slope | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change in urine albumin levels | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change in urine protein levels | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Incidence of changes in echocardiogram results | 12 Months, 24 Months and through study completion (an average of 4.5 years)
  Systolic and diastolic heart function and structure is assessed by ultrasound of the heart. Echocardiogram parameters include left ventricular mass index (LVMi), ejection fraction, fractional shortening, left ventricular mass, valve abnormalities and thickness.
Incidence of changes in Holter ECG | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change of cardiac biomarkers | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Adults only: Response of the heart to external stress induced by exercise measured with Stress test (Bruce protocol) | 12 Months, 24 Months and through study completion (an average of 4.5 years)
  Qualitative evaluation (yes/no) of symptoms (chest pain, shortness of breath, dizziness, palpitations, and other) and the overall impression: normal stress test (yes/no) will be summarized.
  For overall impression only, a shift from baseline will be presented: normal stress test (yes / no).
Adults only: change of Cardiac MRI | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Adults only: change of Brain MRI | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change in plasma level of Gb3 concentration (nM) | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change in plasma level of lyso-Gb3 (nM) | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change in urine level of lyso-Gb3 (nM) | 12 Months, 24 Months and through study completion (an average of 4.5 years)
Change from baseline of Mainz Severity Score Index (MSSI) scores | 12 Months, 24 Months and at the end of study
  Domains (general, neurological, cardiovascular, renal dysfunction)
Incidence of change from baseline in the number of different pain medications | 12 Months, 24 Months and at the end of study
Incidence of Fabry Clinical Events | 12 Months, 24 Months and at the end of study
  FCEs are classified into four categories: renal, cardiac, cerebrovascular and death due to non-cardiac reasons
Adults only: change in Gastrointestinal Symptom Rating Scale (GSRS) scores | 12 Months, 24 Months and at the end of study
  To measure common symptoms of gastrointestinal disorders.
Adults only: change in Brief Pain Inventory - Short Form (BPI-SF) scores | 12 Months, 24 Months and at the end of study
Adults only: change of quality of life assessed using EQ-5D-5L questionnaire | 12 Months, 24 Months and at the end of study
Cohort C only: Change in Gastrointestinal Symptoms (PedsQL-GI) Questionnaire scores | 12 Months, 24 Months and at the end of study
  To measure common symptoms of gastrointestinal disorders.
Cohort C only: change in Fabry-Specific Pediatric Health and Pain Questionnaire (FPHPQ) scores | 12 Months, 24 Months and at the end of study
Cohort C only: change in PedsQL Pediatric Pain Questionnaire (PedsQL-PPQ) scores | 12 Months, 24 Months and at the end of study
Cohort C only: change of quality of life assessed using EQ-5D-Y Questionnaire | 12 Months, 24 Months and at the end of study

CONTACTS AND LOCATIONS:
Locations (9):
- Japan (9):
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Tohoku University Hospital, Sendai, Miyagi
  - University of the Ryukyu Hospital, Nishihara, Okinawa
  - Osaka University Hospital, Suita, Osaka
  - Juntendo University Hospital, 3-1-3 Hongo, Bunkyo-ku, Tokyo, Bunkyo-ku, Tokyo
  - Tokyo Jikei University Hospital, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Asahikawa Medical University Hospital, Asahikawa
  - Niigata University Medical & Dental Hospital, Niigata